CLINICAL TRIAL: NCT01882322
Title: A Phase IV, Randomized, Open-Label, Comparative, Multi-Center Study to Assess the Safety and Efficacy of Advagraf® (Modified Release Tacrolimus, Once Daily) After Using Prograf® (Tacrolimus Twice Daily) in de Novo Liver Transplant Recipients
Brief Title: A Study to Evaluate the Effect of Advagraf Conversion From Prograf in Liver Transplant Subjects
Acronym: Maple
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADV-LT-01
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: de Novo Liver Transplant Subjects
Keywords: FK506; tacrolimus; immunosuppressant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advagraf conversion group (Experimental): Oral
  Interventions: Drug: Prograf; Drug: Advagraf
- Prograf maintenance group (Active Comparator): Oral
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Prograf — oral
  Other Names: Tacrolimus
Drug: Advagraf — oral
  Other Names: modified release Tacrolimus
  Arms: Advagraf conversion group

SUMMARY:
The objective of this study is to compare the efficacy and safety between a group that has been on Prograf twice daily therapy but converted to Advagraf once daily therapy and a group that maintained Prograf twice daily therapy.

DETAILED DESCRIPTION:
De novo Liver Transplant Recipients will be divided into two groups. Both groups will receive Prograf (Tacrolimus twice daily therapy), and at Month 1 (Week 4) after surgery, Prograf will be converted to Advagraf (modified release Tacrolimus, once daily) in one group, while Prograf therapy will be continued in other group.

ELIGIBILITY:
Inclusion Criteria:

* A subject scheduled for liver transplantation from a living donor or brain dead
* In case of a woman of childbearing potential, a subject with a negative pregnancy test prior to enrollment and who consents to and would practice double contraception throughout the study (Pessary therapy, or rhythm method, or sexual abstinence, surgical sterilization, menopause or otherwise sterile; however, oral contraceptives are excluded.)
* A subject with terminal hepatic failure for which liver transplant is necessary
* A subject who understands and is completely aware of the study objective and risks and who submitted a written informed consent form on study participation

Exclusion Criteria:

* A subject who received multiple organ transplants or any previous organ transplant (including re-transplantation of the liver)
* A subject who had received auxiliary transplant or used the bioartificial liver (cellular system)
* A subject allergic or resistant to macrolide antibiotics or Tacrolimus
* A subject who was taking Cyclosporine and Bosentan (Tracleer) that may interact with Tacrolimus, or potassium-sparing diuretics known to possibly cause hyperkalemia (Spironolactone, Triamterene) at screening
* A subject who requires immunosuppressive treatment or systemic chemotherapy from before transplant. However, a subject who received immunosuppressive treatment for less than 1 month prior to transplant to treat underlying hepatic disorder may be enrolled in the study if treatment is discontinued at the time of transplant.
* A subject with malignancy or malignant tumor history within the past 5 years; however, a subject may be enrolled in this study in case of successfully cured for basal cell carcinoma or squamous cell carcinoma of the skin.
* A subject who suffers severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect Tacrolimus absorption (may be determined at the discretion of the investigator)
* A subject with any type of substance abuse, psychological disorder, or communication disorder at the discretion of the investigator
* A subject who is participating in another study or participated within 28 days of the study, or who had received IP or non-registered medication
* A subject who is pregnant or breastfeeding
* A subject (transplant recipient) and/or donor who are positive to HIV
* A subject who cannot comply with the protocol-planned routine visit schedule
* A subject who is not appropriate for study participation at the discretion of the investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01-30 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection | from Week 4 to Week 24 post-transplant
  Acute rejection incidence (%) = Number of subjects with at least one biopsy -confirmed acute rejection / Total number of subjects included in the relevant analysis set * 100

SECONDARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection | from Week 4 to Week 12 or Week 24
Severity of biopsy-confirmed acute rejection | from Week 4 to Week 12 and Week 24 after liver transplant
  Severity guideline is Banff criteria
Subject survival rate and graft survival rate | from Week 4 to Week 12 and Week 24 after liver transplant
Safety assessed by the incidence of adverse events, vital signs, physical exam. and labo-tests | for 24 weeks after liver transplant

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=235